CLINICAL TRIAL: NCT04455464
Title: Effect of Midodrine on HVPG in Advanced Chronic Liver Disease - A Pilot Study
Brief Title: Effect of Midodrine on HVPG in Advanced Chronic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-33
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-10

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midodrine (Experimental): Midodrine will be given 10 mg for one time only. HVPG will be done at baseline and after 3 hours
  Interventions: Drug: Midodrine Oral Tablet

INTERVENTIONS:
Drug: Midodrine Oral Tablet — Midodrine will be given 10 mg for one time only.

SUMMARY:
* Primary objective: HVPG response after administration of midodrine as defined by decrease in HVPG by > 20 % from baseline or to less than equals to 12 mmHg.
* Secondary objectives: Change in HVPG, SVR, heart rate, cardiac output, cardiac index, Blood pressure (systolic, diastolic and mean).

Methodology:

Consecutive patients of chronic liver disease in the Institute (admitted or coming to OPD) as per the inclusion and exclusion criteria will be studied.

* Study Population: Patients of advanced chronic liver disease admitted or OPD patients in ILBS
* Study Design: A single arm interventional study
* Study Period: 6 months
* Inclusion Criteria: i) CLD with grade III ascites with Na < 130 / Systolic BP < 90 / type 2 HRS(n=30 ) (ii) ACLF (APASL criteria) with Na < 130 / Systolic BP < 90 / AKI (n=30)
* Exclusion Criteria: age < 18 and > 75, pregnancy, splanchnic venous thrombosis, HCC, HE, significant cardiopulmonary disease, uncontrolled diabetes, hypertension, intrinsic renal disease, peripheral vascular disease.
* Sample Size with justification: This is a pilot study where a total of 60 patients will be enrolled - 30 each in the two groups.
* Intervention: HVPG will be done in these patients at baseline and then after 3 hours of 10 mg of midodrine tablets.

Monitoring and assessment: Various parameters will be assessed during the procedure before and after 3 hours of midodrine such as HVPG (WHVP - FHVP), SVR, heart rate, cardiac output, cardiac index, Blood pressure (systolic, diastolic and mean), SpO2.

- Statistical Analysis: Continuous data will be represented by mean ± SD or median ± IQR. Categorical data will be represented by n = frequency (%). Categorical data will be analyzed by Chi square test or Fisher exact test as appropriate. Continuous data will be compared by using student t test or Mann Whitney test (when applicable). The change in HVPG will be analyzed by using paired t test or Wilcoxon signed rank test. The % change in the individual group will be compared to see the significance between the groups. The significance will be seen at 5%.

* Adverse Effects: same as for HVPG (mild pain / hematoma at the puncture site, transient arrhythmias). Midodrine has got good safety profile and is used in patients of advanced chronic liver disease.
* Stopping Rule of study: nil

Expected outcome of the project: If result shows that HVPG is decreased by midodrine, then it can be used in place of beta blockers when they are contraindicated or have the potential of causing adverse effects.

ELIGIBILITY:
Inclusion Criteria:

- i) CLD with grade III ascites with Na < 130 / Systolic BP < 90 / type 2 HRS(n=30 ) ii) ACLF (APASL criteria) with Na < 130 / Systolic BP < 90 / AKI (n=30)

Exclusion Criteria:

1. age < 18 and > 75,
2. Pregnancy,
3. Splanchnic venous thrombosis,
4. Hepatocellular Carcinoma,
5. Hepaticencephalopathy,
6. Significant cardiopulmonary disease,
7. Uncontrolled diabetes,
8. Hypertension,
9. Intrinsic renal disease,
10. Peripheral vascular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
HVPG response after administration of midodrine as defined by decrease in HVPG by > 20 % from baseline or to less than equals to 12 mmHg | 3 hours

SECONDARY OUTCOMES:
Change in Hepatic Venous Pressure Gradient. | 3 hours
Change in Systemic Vascular Resistance. | 3 hours
Change in Heart Rate. | 3 hours
Change in Cardiac Output. | 3 hours
Change in Blood pressure (Systolic, Diastolic and Mean). | 3 hours
Change in Cardiac Index. | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided